CLINICAL TRIAL: NCT01940809
Title: A Sequential Safety and Biomarker Study of BRAF-MEK Inhibition on the Immune Response in the Context of Combined CTLA-4 Blockade and PD-1 Blockade for BRAF Mutant Melanoma
Brief Title: Ipilimumab With or Without Dabrafenib, Trametinib, and/or Nivolumab in Treating Patients With Melanoma That Is Metastatic or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01703; NCI-2013-01703 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-304; 9377 (Other: Dana-Farber Cancer Institute); 9377 (Other: CTEP); P30CA006516 (NIH); U01CA062490 (NIH); UM1CA186709 (NIH); NCT01938703 (obsolete NCT alias)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: BRAF V600E Mutation Present; BRAF V600K Mutation Present; Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; Ipilimumab; CTLA-4 Antigen; Nivolumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Arm A1 (ipilimumab, dabrafenib, trametinib) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD for 25 days. Patients then receive ipilimumab IV over 90 minutes. Treatment with ipilimumab repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Arm A2 (dabrafenib, trametinib, nivolumab, ipilimumab) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD for 25 days followed by nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.
  Interventions: Drug: Dabrafenib; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Trametinib
- Arm B1 (ipilimumab, trametinib) (Experimental): Patients receive trametinib PO QD for 25 days. Patients then receive ipilimumab IV over 90 minutes. Treatment with ipilimumab repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Arm B2 (trametinib, nivolumab, ipilimumab) (Experimental): Patients receive trametinib PO QD for 25 days followed by nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Trametinib
- Arm C1 (ipilimumab, dabrafenib) (Experimental): Patients receive dabrafenib PO BID for 25 days. Patients then receive ipilimumab IV over 90 minutes. Treatment with ipilimumab repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis
- Arm C2 (dabrafenib, nivolumab, ipilimumab) (Experimental): Patients receive dabrafenib PO BID for 25 days followed by nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.
  Interventions: Drug: Dabrafenib; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Arm D1 (ipilimumab) (Experimental): Patients receive ipilimumab IV over 90 minutes Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis
- Arm D2 (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
  Arms: Arm A1 (ipilimumab, dabrafenib, trametinib); Arm A2 (dabrafenib, trametinib, nivolumab, ipilimumab); Arm C1 (ipilimumab, dabrafenib); Arm C2 (dabrafenib, nivolumab, ipilimumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: Arm A2 (dabrafenib, trametinib, nivolumab, ipilimumab); Arm B2 (trametinib, nivolumab, ipilimumab); Arm C2 (dabrafenib, nivolumab, ipilimumab); Arm D2 (nivolumab, ipilimumab)
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212
  Arms: Arm A1 (ipilimumab, dabrafenib, trametinib); Arm A2 (dabrafenib, trametinib, nivolumab, ipilimumab); Arm B1 (ipilimumab, trametinib); Arm B2 (trametinib, nivolumab, ipilimumab)

SUMMARY:
This randomized phase I trial studies the side effects and best way to give ipilimumab with or without dabrafenib, trametinib and/or nivolumab in treating patients with melanoma that has spread to other parts of the body (metastatic) or cannot be removed by surgery. Monoclonal antibodies, such as ipilimumab and nivolumab, may interfere with the ability of cancer cells to grow and spread. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether ipilimumab works better with or without dabrafenib, trametinib, and/or nivolumab in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of ipilimumab (part 1) or ipilimumab plus nivolumab (part 2) following lead-in of v-raf murine sarcoma viral oncogene homolog B1 (BRAF) and mitogen-activated protein kinase kinase (MEK) inhibitors, either alone or in combination, in patients with BRAFV600 mutant melanoma.

SECONDARY OBJECTIVES:

I. To determine the response rate to ipilimumab (part 1) or ipilimumab plus nivolumab (part 2) after BRAF and MEK inhibitors, either alone or in combination, compared to no prior kinase inhibitor treatment.

II. To determine the safety and tolerability of dabrafenib and trametinib combination in the setting of prior ipilimumab alone or ipilimumab preceded by BRAF and MEK inhibitors, either alone or in combination (part 1).

III. To determine the safety and tolerability of dabrafenib and trametinib combination in the setting of prior ipilimumab plus nivolumab without prior BRAF/MEK inhibition or ipilimumab plus nivolumab preceded by BRAF and MEK inhibitors, either alone or in combination (part 2).

IV. To determine the response rate to dabrafenib and trametinib in the setting of prior ipilimumab alone or ipilimumab preceded by BRAF and MEK inhibitors, either alone or in combination (part 1).

V. To determine the response rate to dabrafenib and trametinib in the setting of prior ipilimumab plus nivolumab without prior MEK/BRAF inhibition or prior ipilimumab plus nivolumab preceded by BRAF/MEK inhibitors (part 2).

VI. To obtain peripheral blood and tumor tissue for biomarker analysis. VII. To describe the immune impact of kinase inhibitor therapy on the immune response associated with ipilimumab treatment (part 1) or ipilimumab plus nivolumab treatment (part 2).

VIII. To observe and record anti-tumor activity.

OUTLINE: Patients are randomized to 1 of 4 treatment arms for Part 2 (Part 1 closed to accrual 8/25/2015).

PART 1: (Closed to accrual as of 8/25/2015) ARM A1: Patients receive dabrafenib orally (PO) twice daily (BID) and trametinib PO once daily (QD) for 25 days. Patients then receive ipilimumab intravenously (IV) over 90 minutes. Treatment with ipilimumab repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM B1: Patients receive trametinib PO QD for 25 days. Patients then receive ipilimumab IV over 90 minutes. Treatment with ipilimumab repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM C1: Patients receive dabrafenib PO BID for 25 days. Patients then receive ipilimumab IV over 90 minutes. Treatment with ipilimumab repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM D1: Patients receive ipilimumab IV over 90 minutes. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

PART 2:

ARM A2: Patients receive dabrafenib PO BID and trametinib PO QD for 25 days followed by nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.

ARM B2: Patients receive trametinib PO QD for 25 days followed by nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.

ARM C2: Patients receive dabrafenib PO BID for 25 days followed by nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.

ARM D2: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 4 doses, followed by nivolumab monotherapy IV every 2 weeks continuously for up to 42 courses.

After 12 weeks of treatment with ipilimumab, or ipilimumab and nivolumab followed by nivolumab monotherapy, all patients may continue to receive dabrafenib PO BID and trametinib PO QD in the absence of disease progression.

After completion of study treatment, patients are followed up for 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have histologically or cytologically confirmed unresectable or metastatic malignant melanoma
* Study participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Study participants must have completed any prior treatment at least 3 weeks prior to treatment on this protocol; prior treatments may have included chemotherapy however may not have included BRAF or MEK inhibitors or immunotherapies (interleukin-2, ipilimumab, anti-programmed death [PD]1 antibodies etc.) excluding vaccine therapy; prior treatment with interferon in the adjuvant setting is allowed, though prior treatment with ipilimumab in the adjuvant setting is not; prior radiation therapy is allowed though must have included no more than 3000 centigray (cGy) to fields including substantial marrow
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1.2 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Albumin >= 2.5 g/dL
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) except subjects with known Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.3 x institutional ULN; subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to randomization
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO)
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Patients must have BRAFV600E or BRAFV600K mutations, identified by a Food and Drug Administration (FDA)-approved test at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory (lab); if test at CLIA-certified lab used a non-FDA approved method, information about the assay must be provided
* Therapeutic level dosing of warfarin can be used with close monitoring of PT/INR by the site; exposure may be decreased due to enzyme induction when on treatment, thus warfarin dosing may need to be adjusted based upon PT/INR; consequently, when discontinuing dabrafenib, warfarin exposure may be increased and thus close monitoring via PT/INR and warfarin dose adjustments must be made as clinically appropriate; prophylactic low dose warfarin may be given to maintain central catheter patency
* Women of child-bearing potential must agree to use adequate contraception (barrier method of birth control, or abstinence; hormonal contraception is not allowed) for the duration of study participation, and for at least 2 weeks after treatment with dabrafenib or for 6 months after dabrafenib in combination with trametinib; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 grade =< 1 (except alopecia) at the time of randomization
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior systemic anti-cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or vaccine therapy) within the last 3 weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks preceding the first dose of study treatment
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study treatment and during the study
* Study participants with a history of prior treatment with BRAF or MEK inhibitors
* Study participants who had prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible

  * Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Study participants who have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Study participants with known immune impairment who may be unable to respond to anti-cytotoxic T-lymphocyte antigen 4 (CTLA 4) antibody and/or anti-PD-1 antibody
* Study participants with brain metastases are excluded unless these have been definitively treated and are radiographically stable for at least 1 month; the study participant must also demonstrate a stable physical exam and must have discontinued systemic steroids for treatment of edema related to brain metastases or treatment for over 7 days
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* Current use of a prohibited medication; patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A (CYP3A) or cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) are ineligible; current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* A history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (with the exception of cleared HBV and HCV infection, which will be allowed)
* Patients with history of rat sarcoma (RAS) mutation-positive tumors are not eligible regardless of interval from the current study; Note: prospective RAS testing is not required; however, if the results of previous RAS testing are known, they must be used in assessing eligibility
* History or evidence of cardiovascular risks including any of the following:

  * QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within the past 24 weeks prior to randomization
  * History or evidence of current class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Intra-cardiac defibrillators
  * Abnormal cardiac valve morphology (>= grade 2) documented by ECHO; (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study); subjects with moderate valvular thickening should not be entered on study
  * History or evidence of current clinically significant uncontrolled cardiac arrhythmias; clarification: subjects with atrial fibrillation controlled for > 30 days prior to dosing are eligible
  * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation
* History of retinal vein occlusion (RVO)
* History of interstitial lung disease or pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher immune-related adverse events (irAEs), graded according to the National Cancer Institute (NCI) CTCAE v4.0 | Up to 3 weeks after end of ipilimumab induction
  Presented with 90% confidence intervals calculated using exact binomial methods.

SECONDARY OUTCOMES:
Proportion of patients receiving dabrafenib and trametinib with grade 3 or higher irAEs after disease progression on ipilimumab, according to the NCI CTCAE v4.0 | Up to 4 weeks after completion of study treatment
  Presented with 90% confidence intervals calculated using exact binomial methods by randomized treatment arm.
Response rate for the total treatment period according to Response Evaluation Criteria in Solid Tumors v1.1 | Up to 4 weeks after completion of study treatment
  Summarized by treatment arm and presented with 90% exact binomial confidence intervals. Fisher's exact test will be used.
Disease-control rate | Up to 4 weeks after completion of study treatment
  Summarized by treatment arm and presented with 90% exact binomial confidence intervals. Fisher's exact test will be used.

OTHER OUTCOMES:
Biomarker expression levels | Baseline
  The relationship between pre-treatment marker levels and response will be assessed according to expression cut-off between positive and negative. Fisher's exact test will be used to detect an increase in response rate and a secondary, sensitivity analysis will use a stratified Fisher's exact test.
Fold-changes in biomarkers | Baseline to 3 weeks after fourth ipilimumab dose
  Biomarkers measured on a continuous scale will be summarized and compared across response categories using the Wilcoxon rank-sum test. For biomarkers measured categorically, pre/post response combinations will be compared between responders and non-responders using Fisher's exact test.
Change in immune activation, measured by changes in biomarker levels | Baseline to 3 weeks after fourth ipilimumab dose
  Biomarkers measured on a continuous scale will be summarized and compared across response categories using the Wilcoxon rank-sum test. For biomarkers measured categorically, pre/post response combinations will be compared between responders and non-responders using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Ott, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts